CLINICAL TRIAL: NCT04365530
Title: Become of Patients Infected or Suspected of Being Infected by Covid-19 and Supported by the GHPSJ and the Establishments of the Paris Plaisance Hospital City
Acronym: COVIDGHPSJCite
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Cohorte COVID GHPSJ CiteH
Record Dates: First submitted 2020-04-26; First posted 2020-04-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ongoing Coronavirus (Covid-19) pandemic is causing a major global health crisis and is shaking up hospital organizations. To date, the recognized risk factors for severe forms of Covid-19 infection are elderly patients (> 70 years), obese patients, patients with chronic renal or respiratory pathologies, cardiovascular history (stroke or coronary artery disease), chronic respiratory conditions, high blood pressure, diabetes, and cancer. Covid-19 is manifested by a risk of acute respiratory distress syndrome requiring management by invasive ventilation. The lethality of this infection is around 4% in the current data.

Drastic precautionary measures for the transmission of the virus, as well as the provision of critical care beds by canceling any scheduled non-urgent intervention or consultation, have shaken up the hospital organization.

In this context, it is essential to have forward-looking data in real time to adjust the care offer and better understand the impact of Covid-19 on the patient populations treated.

ELIGIBILITY:
Inclusion Criteria:

- Patient (of all ages) with symptoms compatible with infection by Covid-19 treated at the GHPSJ or in one of the establishments in the Paris Plaisance hospital city.

Exclusion Criteria:

* Asymptomatic patient
* Patient objecting to the use of their data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patientwith symptoms compatible with infection by Covid-19 treated at the GHPSJ or in one of the establishments in the Paris Plaisance hospital city.
Sampling Method: Non-Probability Sample
Enrollment: 3767 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Clinical consequences of a Covid-19 infection in the care population | Year 2
  This outcome measures the clinical consequences of a Covid-19 infection in the care population.

SECONDARY OUTCOMES:
Risk factors at M6 | Month 6
  This outcome evaluates the risk factors of COVID-19 at month 6
Risk factors at year 1 | Year 1
  This outcome evaluates the risk factors of COVID-19.
Risk factors at year 2 | Year 2
  This outcome evaluates the risk factors of COVID-19.
Impact of hospital reorganization on medical care at M6 | Month 6
  This outcome evaluates the impact of hospital reorganization on medical care at month 6.
Impact of hospital reorganization on medical care at Year 1 | Year 1
  This outcome evaluates the impact of hospital reorganization on medical care at year 1.
Impact of hospital reorganization on medical care at Year 2 | Year 2
  This outcome evaluates the impact of hospital reorganization on medical care at year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (5):
- France (5):
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - AURA Paris Plaisance, Paris
  - Fondation Sainte-Marie, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hôpital Bellan, Paris